CLINICAL TRIAL: NCT01093521
Title: A Pharmacokinetic and Safety Study of IV Gallium Nitrate (Ganite) in Cystic Fibrosis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Chris Goss, Associate Professor, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 35876; US FDA 5R01FD003704 (Other Grant/Funding Number: FDA)
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Results first posted 2016-01-12 (Estimated); Last update posted 2022-11-29 (Actual); Status verified 2022-10

CONDITIONS: Cystic Fibrosis
Keywords: IV Gallium; Gallium; Ganite; Cystic Fibrosis; Gallium Infusion
MeSH Terms: conditions — Cystic Fibrosis | interventions — gallium nitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 100 mg/m2 dose (Experimental): Five day continuous IV Gallium Nitrate (Ganite®) infusion at 100 mg/m2
  Interventions: Drug: 100 mg/m2 dose
- 200 mg/m2 dose (Experimental): Five day continuous IV Gallium Nitrate (Ganite®) infusion at 200 mg/m2
  Interventions: Drug: 200 mg/m2 dose

INTERVENTIONS:
Drug: 100 mg/m2 dose — 5 day infusion of gallium nitrate (IV Ganite®) at a dose of 100 mg/m2/day
  Other Names: Ganite®; gallium nitrate
  Arms: 100 mg/m2 dose
Drug: 200 mg/m2 dose — 5 day infusion of gallium nitrate (IV Ganite®) at 200 mg/m2/day
  Other Names: Ganite®; gallium nitrate
  Arms: 200 mg/m2 dose

SUMMARY:
The purpose of this research study is to test the pharmacokinetics, safety, and tolerability of an intravenous infusion of a drug called Ganite (gallium nitrate) in patients with cystic fibrosis. We want to see this drug is safe and tolerable and to see if high levels of the drug are found in the sputum.

Funding Source - Food and Drug Administration (FDA) Office of Orphan Products Development (OOPD)

DETAILED DESCRIPTION:
This is a two center pharmacokinetic and safety dosing study of IV gallium nitrate (Ganite®) in cystic fibrosis (CF) patients. Eighteen subjects are planned. Each subject will be administered a single 5-day infusion of study medication (one of 2 doses). No placebo is used. Each subject will receive 5 days of continuous infusion of the experimental treatment. There will be two dosing cohorts (cohort 1: 100 mg/m2/day and cohort 2: 200 mg/m2/day). Cohort 2 will begin enrollment only after Data Safety Monitoring Committee (DSMC) safety review and approval of cohort 1 data. Study visits occur at baseline (day 1), day 3 (visit 2), day 6 (visit 3), day 8 (visit 4), day 14 (visit 5), day 28 (visit 6), and day 56 (visit 7).

Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study.

The following treatment regimens will be used:

• Experimental treatment continuous infusion of gallium nitrate at the following doses cohort 1: 100 mg/m2/day and cohort 2: 200 mg/m2/day All subjects who receive at least one dose of study medication will be considered evaluable for safety and efficacy analyses. Incidence of adverse events will be monitored during the trial.

Primary endpoints will be assessment of pharmacokinetic and safety/tolerability data.

Secondary efficacy assessments will be based on changes in lung function and sputum P. aeruginosa density in sputum.

Total duration of subject participation will be five weeks. Total duration of the study is expected to be 20 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female, between 18 and 55 years of age
2. Documented chronic colonization with Pseudomonas Aeruginosa (Pa)
3. Confirmed diagnosis of CF:

   1. Documented history of > 60 mmol/L chloride concentration in pilocarpine sweat chloride test And/Or
   2. Genotype with two identifiable mutations consistent with CF, accompanied by one or more phenotypic features consistent with diagnosis of CF
4. Forced expiratory volume in the first second (FEV1) ≥ 30% of predicted value
5. Able to expectorate sputum
6. Serum liver function tests ≤ 2.5 x upper limit of normal
7. Serum urea nitrogen (BUN) and creatinine ≤ 1.5 x upper limit of normal
8. Serum creatinine ≤ 2.0 mg/dl
9. Hemoglobin ≥ 9 g/dl, platelets ≥ 100,000/mm3, and white blood cells (WBC) ≥ 4,500/mm3 and ≤ 15,000/mm3
10. Ionized calcium ≥ the lower limit of normal
11. Able to understand and sign the informed consent document, communicate with the Investigator, and comply with the requirements of the protocol
12. If female and of childbearing potential, must have a negative pregnancy test on Day 1 prior to receiving study drug
13. If female and of childbearing potential, is willing to use adequate contraception, as determined by the investigator, for the duration of the study

Exclusion Criteria:

1. Acute pulmonary exacerbation requiring antibiotic intervention within 2 weeks prior to screening
2. Osteoporosis defined as the most recent dexa scan within the prior 5 years with a T-score ≤ -2.5
3. Pregnant or lactating female
4. Known sensitivity to gallium
5. Use of biphosphonates
6. Use of any investigational drug and/or participated in any clinical trial within 3 months prior to screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2012-04 (Actual); Study Completion 2013-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher H Goss, MD, MSc, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in the Adult cystic fibrosis clinics at 3 centers (the University of Washington, University of Iowa, John's Hopkins University) from the second quarter 2010 and closed February 1, 2012. The study had two dosing cohorts. Cohort 1 completed enrollment in February, 2011. Cohort 2 completed enrollment on February 1, 2012.
Pre-assignment Details: We employed no run-in period. No subjects withdrew after randomization.
Groups:
- IV Gallium (Ganite®) Infusion: Five day continuous IV Gallium (Ganite®)infusion
  IV Gallium Nitrate (Ganite®) infusion: 5 day infusion of gallium nitrate (IV Ganite®) at a doses of 100 mg/m2/day and 200 mg/m2/day and 5 day infusion of gallium nitrate (IV Ganite®) 100 mg/m2/day and 200 mg/m2/day
Period: Overall Study
Arm/Group | IV Gallium (Ganite®) Infusion
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients were adults age 18 years but less than 55 years of age with CF and chronic Pseudomonal infection. Patient had to have a baseline FEV1% of predicted greater than or equal to 30%. They had to have been at least 14 days from the end of treatment with intravenous antibiotics for exacerbation. They could not be lactating or pregnant.
Arm/Group | IV Gallium (Ganite®) Infusion
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 20
Forced expiratory volume in one second (FEV1) (in liters) [Mean (Full Range); unit: liters] | 2.25 [1.06 to 4.59]
Forced vital capacity (FVC)(in liters) [Mean (Full Range); unit: liters] | 3.60 [1.84 to 6.11]
Mean Pseudomonas aeruginosa quantitative sputum culture (CFU's/gr of sputum) [Mean (Full Range); unit: Million CFU/gr of sputum] | 116.7 [0.378 to 866]

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Assessment of a 5 Day Infusion of Gallium Nitrate (IV Ganite®)
Description: To assess the summed area under the curves of a 5 day infusion of IV Ga from day 1 to day 28 at two doses: 100 mg/m2/day in adult subjects with CF; 200 mg/m2/day in adult subjects with CF.
  To assess the safety of a 5 day infusion of IV Ga at two doses: 100 mg/m2/day in adult subjects with CF; 200 mg/m2/day in adult subjects with CF.
  Safety and tolerability of 5 days of treatment with IV administered gallium nitrate (IV Ganite®) at a doses of 100 mg/m2/day and 200 mg/m2/day.
Time Frame: Day 1 at t=1, 2 and 6 hours, Day 3, Day 6 at t= 1, 2, 8, and 12, Day 14 and Day 28
Measure: Mean (Standard Deviation); unit: ug*hr/mL
Groups:
- IV Gallium (Ganite®) Infusion 100 mg/m2/Day: Five day continuous IV Gallium (Ganite®)infusion
  IV Gallium Nitrate (Ganite®) infusion: 5 day infusion of gallium nitrate (IV Ganite®) at a doses of 100 mg/m2/day
- IV Gallium (Ganite®) Infusion 200 mg/m2/Day: Five day continuous IV Gallium (Ganite®)infusion
  IV Gallium Nitrate (Ganite®) infusion: 5 day infusion of gallium nitrate (IV Ganite®) at a doses of 200 mg/m2/day
Arm/Group | IV Gallium (Ganite®) Infusion 100 mg/m2/Day | IV Gallium (Ganite®) Infusion 200 mg/m2/Day
Number analyzed (Participants) | 9 | 11
ug*hr/mL | 503 (98) | 537 (153)

2. Secondary Outcome: Change in Spirometry From Baseline to Day 8
Description: Change in spirometry as measured by FEV1 in liters from baseline to day 8
Time Frame: 8 days
Population: ITT
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | IV Gallium (Ganite®) Infusion
Number analyzed (Participants) | 20
liters | 0.13 (0.18)

3. Secondary Outcome: Change in Lung Function From Baseline to Day 15
Description: Change in FEV1 in liters from baseline to day 15
Time Frame: 15 days from starting dose
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | IV Gallium (Ganite®) Infusion
Number analyzed (Participants) | 20
liters | 0.13 (0.17)

4. Secondary Outcome: Change in Spirometry From Baseline to Day 28
Description: Change in lung function as measured by FEV1 in liters from baseline to day 28
Time Frame: 28 days from starting dose
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | IV Gallium (Ganite®) Infusion
Number analyzed (Participants) | 20
liters | 0.10 (0.14)

5. Secondary Outcome: Change in Spirometry From Baseline to Day 56
Description: Change in lung function as measured by FEV1 in liters from baseline to day 56
Time Frame: 56 days from starting dose
Population: all those subjects enrolled after the amendment to add a day 56 (ITT)
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | IV Gallium (Ganite®) Infusion
Number analyzed (Participants) | 11
liters | 0.12 (0.19)

6. Secondary Outcome: Change in Spirometry as Measured by FVC From Baseline to Day 8
Description: Change from baseline in lung function assessed by FVC in liters after treatment with IV Ga at day 8
Time Frame: 8 days from starting dose
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | IV Gallium (Ganite®) Infusion
Number analyzed (Participants) | 20
liters | 0.16 (0.20)

7. Secondary Outcome: Change in P. Aeruginosa Density From Baseline to Day 8
Description: Change in sputum microbiology (specifically P. aeruginosa density based on quantitative cultures) from baseline to day 8
Time Frame: 8 days from starting dose
Population: All available specimens
Measure: Mean (Standard Deviation); unit: colony counts in millions per gm sputum
Arm/Group | IV Gallium (Ganite®) Infusion
Number analyzed (Participants) | 19
colony counts in millions per gm sputum | 21.1 (297.5)

8. Secondary Outcome: Change in Sputum P. Aeruginosa Density From Baseline to Day 15
Description: Change in sputum microbiology (specifically P. aeruginosa density based on quantitative cultures) from baseline to day 15
Time Frame: 15 days from starting dose
Measure: Mean (Standard Deviation); unit: colony counts in millions per gm sputum
Arm/Group | IV Gallium (Ganite®) Infusion
Number analyzed (Participants) | 19
colony counts in millions per gm sputum | -5.5 (217.9)

9. Secondary Outcome: Change in P. Aeruginosa Density From Baseline to Day 56
Description: Change in sputum microbiology (specifically P. aeruginosa density based on quantitative cultures) from baseline to day 56
Time Frame: 56 days from starting dose
Population: All available specimens
Measure: Mean (Standard Deviation); unit: colony counts in millions per gm sputum
Arm/Group | IV Gallium (Ganite®) Infusion
Number analyzed (Participants) | 5
colony counts in millions per gm sputum | -76.0 (58.3)

10. Primary Outcome: Number of Serious Adverse Events
Description: Safety as measured by serous adverse events
Time Frame: 56 days from starting dose
Population: ITT
Measure: Number; unit: Serious Adverse Events
Arm/Group | IV Gallium (Ganite®) Infusion
Number analyzed (Participants) | 20
Serious Adverse Events | 0

11. Primary Outcome: Number of Events When Study Drug Infusion Was Stopped Early
Description: Tolerability as measured by adverse events of a 5 day continuous infusion of IV Gallium as assessed by stopping study drug infusion
Time Frame: 6 days from starting dose
Measure: Number; unit: Number of times study drug interupted
Arm/Group | IV Gallium (Ganite®) Infusion
Number analyzed (Participants) | 20
Number of times study drug interupted | 0

ADVERSE EVENTS:
Time Frame: 56 days
Description: At study visits, all body systems were assessed for adverse events. Serious adverse events were assessed at all study visits and participants were told to inform their research team of any serious adverse events occurring between study visits.
Arm/Group | IV Gallium (Ganite®) Infusion
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 18/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Gallium (Ganite®) Infusion (N=20)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) — Lymphadenopathy
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 3 (3) — Cystic fibrosis lung exacerbation
External ear inflammation (Ear and labyrinth disorders) | 2 (2) — otitis externa
Abdominal distension (Gastrointestinal disorders) | 1 (1) — Abdominal distension
Abdominal pain (Gastrointestinal disorders) | 2 (2) — Abdominal pain
Gastrointestinal reflux disease (Gastrointestinal disorders) | 1 (1) — Gastrointestinal reflux disease
Nausea (Gastrointestinal disorders) | 1 (1) — Nausea
Stomach discomfort (Gastrointestinal disorders) | 1 (1) — Stomach discomfort
vomiting (Gastrointestinal disorders) | 1 (1) — vomiting
fatigue (General disorders) | 4 (4) — fatigue
Peripheral edema (General disorders) | 1 (1) — peripheral edema
pyrexia (General disorders) | 1 (1) — fever
urinary tract infection (Infections and infestations) | 1 (5) — urinary tract infection
infusion site bruising (Injury, poisoning and procedural complications) | 3 (3) — infusion site bruising
infusion site hematoma (Injury, poisoning and procedural complications) | 1 (1) — infusion site hematoma
infusion site pain (Injury, poisoning and procedural complications) | 1 (1) — infusion site pain
infusion site swelling (Injury, poisoning and procedural complications) | 1 (1) — infusion site swelling
Blood glucose increased (Investigations) | 1 (1) — increased blood glucose
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) — Back pain
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) — Gout
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) — Muscle spasms
neck stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) — Neck stiffness
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) — Pain in extremity
Dizziness (Nervous system disorders) | 1 (1) — dizziness
headache (Nervous system disorders) | 9 (16) — headache
Migraine (Nervous system disorders) | 1 (1) — Migraine headache
Paresthesia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
albuminuria (Renal and urinary disorders) | 1 (1) — albuminuria
Haematuria (Renal and urinary disorders) | 2 (2)
Pyuria (Renal and urinary disorders) | 1 (1) — Pyuria
Pelvic pain (Reproductive system and breast disorders) | 1 (1) — Pelvic pain
cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) — increased cough
crackles lung (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Crackles heard on lung exam
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Dyspnoea
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (5) — Haemoptysis
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Nasal congestion
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Epistaxis
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Non-cardiac chest pain
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Productive cough
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) — rhinitis
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) — sinus congestion
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Sinus disorder
Sputum discolored (Respiratory, thoracic and mediastinal disorders) | 1 (1) — sputum discolored
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Throat irritation
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Upper respiratory tract infection
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Voice alteration
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Rash

LIMITATIONS AND CAVEATS:
The primary limitation of our study was that it was uncontrolled without a blinded placebo. Thus, subjective endpoints could have been biased by either the subjects or the investigators.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No